CLINICAL TRIAL: NCT05148936
Title: Communities Fighting COVID!
Brief Title: Communities Fighting COVID-19!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan M Kiene, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-2020-0186; 3U54CA132384-10S1 (NIH)
Record Dates: First submitted 2021-03-31; First posted 2021-12-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- At home testing (Aim 1) (Experimental): High-risk friends and family of contacts exposed to COVID-19 will be provided with COVID-19 testing provided at home by a healthcare worker.
  Interventions: Other: COVID-19 Testing Home-based (Aim 1)
- Mobile testing (Aim 1) (Active Comparator): High-risk friends and family of contacts exposed to COVID-19 will be referred to study operated mobile testing sites in the community for COVID-19 testing.
  Interventions: Other: COVID-19 Testing Mobile (Aim 1)
- Mobile testing approach 1 (Aim 2) (Other): Mobile testing utilizing active outreach
  Interventions: Other: COVID-19 Testing Mobile Approach 1 (Aim 2)
- Mobile testing approach 2 (Aim 2) (Other): Mobile testing utilizing baseline outreach approaches
  Interventions: Other: COVID-19 Testing Mobile Approach 2 (Aim 2)

INTERVENTIONS:
Other: COVID-19 Testing Home-based (Aim 1) — Implementation of Antigen and PCR testing at participant homes
  Arms: At home testing (Aim 1)
Other: COVID-19 Testing Mobile (Aim 1) — Implementation of Antigen and PCR testing at mobile test sites
  Arms: Mobile testing (Aim 1)
Other: COVID-19 Testing Mobile Approach 1 (Aim 2) — Implementation of Antigen and PCR testing at mobile test sites - active outreach
  Arms: Mobile testing approach 1 (Aim 2)
Other: COVID-19 Testing Mobile Approach 2 (Aim 2) — Implementation of Antigen and PCR testing at mobile test sites - baseline outreach
  Arms: Mobile testing approach 2 (Aim 2)

SUMMARY:
To create and evaluate effective COVID-19 testing uptake strategies that focus on underserved individuals who are exposed but have not accessed testing, and underserved individuals who are not routinely tested because they are unaware of their exposure or risk status in order to increase testing among these populations and reduce Covid-19 related disparities.

DETAILED DESCRIPTION:
Communities Fighting COVID is a partnership between San Diego State's School of Public Health and numerous communities in San Diego focused on providing community-based testing to specific language-speaking communities and vulnerable populations. This partnership is funded by the National Institutes of Health (NIH) Rapid Acceleration of Diagnostics-Undeserved Populations (Radx-UP), with the aim of ensuring all Americans have access to timely COVID-19 testing and diagnosis. Many communities, particularly immigrant and people of color communities, have a harder time accessing existing COVID-19 resources due to transportation, language barriers, or other barriers.

ELIGIBILITY:
Inclusion Criteria:

* African American, Arabic speaking, Filipino, and Latino/a populations

Exclusion Criteria:

* Younger than 6, not in focus populations

Ages: 6 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32750 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Test uptake | Through study completion, expected to be 20 months
  Testing volume by study arm as cumulative count per hours testing site operated

SECONDARY OUTCOMES:
Test access | Through study completion, expected to be 20 months
  Proportion of individuals by study arm who note that this strategy has facilitated ability to test.
Test Impact (COVID-19 diagnoses) | Through study completion, expected to be 20 months
  Proportion of COVID-19 diagnoses of those tested by study arm
Test Impact (number needed to screen) | Through study completion, expected to be 20 months
  Number needed to screen (number tested in order to detect one new infection).

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Kiene, PhD, Principal Investigator — San Diego State University
Locations (1):
- Contact Households, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share with Rad-X UP Coordinating Center
Supporting Information: Study Protocol, SAP
Time Frame: Shared on a periodic basis. RPPR shared with NIH on a 6-month basis
Access Criteria: Anonymized data access